CLINICAL TRIAL: NCT06325462
Title: The Influence of Different Anesthetic Techniques on Cerebral Oxygenation During Spinal Surgery in a Prone Position With Controlled Hypotension
Brief Title: The Influence of Anesthetic Technique on Cerebral Oxygenation During Spinal Surgery
Status: Completed | Type: Observational
Sponsor: Prince Sultan Military Medical City (Other)
Responsible Party: Principal Investigator, Mohamed Daabiss, Principal investigator, Prince Sultan Military Medical City
Other Study IDs: E2232/2023
Record Dates: First submitted 2024-03-09; First posted 2024-03-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Oxygenation
Keywords: prone position; controlled hypotension; cerebral oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group S: 27 patients will receive inhalational general anesthesia using sevoflurane.
  Interventions: Device: sensors of regional cerebral oxygen saturation (O3 regional oximeter, Masimo Corp, Irvine, CA) FDA Reg No. 3011353843
- Group P: 27 patients will receive intravenous anesthesia using propofol infusion.
  Interventions: Device: sensors of regional cerebral oxygen saturation (O3 regional oximeter, Masimo Corp, Irvine, CA) FDA Reg No. 3011353843

INTERVENTIONS:
Device: sensors of regional cerebral oxygen saturation (O3 regional oximeter, Masimo Corp, Irvine, CA) FDA Reg No. 3011353843 — O3 regional oximetry monitors the regional hemoglobin oxygen saturation of the blood (rSO2) in adult patients, placed on the forehead by noninvasive and continuous combining arterial and venous oxygen saturation signals from near-infrared spectroscopy (NIRS)

SUMMARY:
Postural changes during anesthesia can lead to decreased cerebral blood flow and oxygenation, especially when moving from a supine to a prone position. This is particularly relevant during spinal surgery with controlled hypotension. Cerebral oximetry, monitored in the frontal cortex using an O3 sensor, is a noninvasive and continuous method to investigate the impact of anesthetic techniques on cerebral oxygenation in such scenarios.

DETAILED DESCRIPTION:
All patients will be monitored with standard monitoring, SedLine sedation monitor, and O3 regional oximeter, Masimo Corp, Irvine, CA. Fentanyl, propofol, and cisatracurium will be administered for anesthesia induction. Anesthetic agents will be maintained with intravenous anesthetic agents in one group and sevoflurane in another group to obtain the PSI 25-50. Mean blood pressure will be maintained 20-30% below baseline. MAP, HR, SpO2, ETCO2, and SrO2 will be assessed at supine position without oxygen administration (T1), supine position with oxygen administration (T2-baseline), intubation in the supine position (T3), just after prone positioning (T4), 10 minutes after prone positioning (T5), at the end of surgery in the prone position (T6) and at the end of anesthesia in the supine position (T7).

Data will be expressed as mean and standard deviation. The mean differences will be analyzed using the Student's T test for quantitative variables in those cases in which those variables followed a normal distribution. Distribution will be evaluated by Kolmogorov-Smirnoff's Z test. Differences in proportion will be conducted with contingency analysis using Chi-square and Fisher's exact test when needed.

A P-value < 0.05 will be statistically significant. Statistical analysis will be performed using the SPSS-PC statistical software program (version 15.0; SPSS, Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status I and II
* Scheduled for elective spinal surgery
* Prone position
* General anesthesia with controlled hypotension.

Exclusion Criteria:

* Hypertension
* Coronary artery disease
* Renal, hepatic, or cerebral insufficiency,
* Patients with coagulopathy or receiving drugs affecting coagulation
* Grossly anemic
* Hypovolemic patients
* Chronically diseased and debilitated patients,
* Bleeding more than 200 mL
* Hemodynamic instability (decrease of 25% of baseline mean arterial pressure [MAP] for three minutes)
* Patients with significant baseline bradycardia.

Ages: 18 Years to 68 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Fifty-four patients of both sexes between 18 and 68 years
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
regional cerebral oxygen saturation | up to 24 weeks
  By applying the sensors of regional cerebral oxygen saturation on the forehead.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Daabiss, M.D., Principal Investigator — Prince Sultan Military Medical City
Locations (1):
- Prince Sultan Military Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chaix I, Manquat E, Liu N, Casadio MC, Ludes PO, Tantot A, Lopes JP, Touchard C, Mateo J, Mebazaa A, Gayat E, Vallee F. Impact of hypotension on cerebral perfusion during general anesthesia induction: A prospective observational study in adults. Acta Anaesthesiol Scand. 2020 May;64(5):592-601. doi: 10.1111/aas.13537. Epub 2020 Jan 19. PMID 31883375
- See also: Effect of Deliberate Hypotension on Regional Cerebral Oxygen Saturation During Functional Endoscopic Sinus Surgery: A Randomized Controlled Trial — https://www.frontiersin.org/articles/10.3389/fsurg.2021.681471/full